CLINICAL TRIAL: NCT05658588
Title: Impact of Cytosorb and CKRT on Hemodynamics in Pediatric Patients With Septic Shock: the PedCyto Study
Brief Title: Hemodynamic Impact of Cytosorb and CKRT in Children With Septic Shock
Acronym: PedCyto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Pediatrico Bambin Gesù (Other)
Responsible Party: Principal Investigator, Gabriella Bottari, Medical Doctor, Principal Investigator, Pediatric Intensivist, Ospedale Pediatrico Bambin Gesù
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR-GB01
Record Dates: First submitted 2022-12-04; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Septic Shock
Keywords: Pediatric Septic Shock; Blood Purification; AKI; Pediatric Critical Care; Hemoperfusion; CKRT
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: a two-stage plan by Simon
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemoperfusion and CKRT in pediatric septic shock (Experimental): Hemoperfusion with Cytosorb in combination with CKRT
  Interventions: Device: Cytosorb

INTERVENTIONS:
Device: Cytosorb — Cytosorb cartridge It is composed of polystyrene divinylbenzene and polyvinylpyrrolidone copolymers and targets molecules in the 5-50 kDa range, which includes the molecular mass of several cytokines
  Other Names: CKRT

SUMMARY:
Impact of the hemoadsorption with Cytosorb on hemodynamic in pediatric patients with septic shock: a prospectic pediatric pilot study

DETAILED DESCRIPTION:
Prospective interventional pilot study included children with septic shock, weight ≥ 10 Kgs and requiring continuous kidney replacement therapy. Cytosorb (CytoSorbents Inc, New Jersey, USA) cartridge was added to CKRT every 24 hours for a maximum of 96 hours. A control group of matched patients was also identified from an external database. The primary outcome of the study was the proportion of patients who achieved an equal or more than 50% relative reduction in vasopressors or inotropes dose from baseline to the end of treatment. Secondary outcomes included doses of vasopressors and inotropes, hemodynamic and biological changes, changes in severity scores and 28-day mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Children weighing ≥ 10 kg
2. Septic shock as defined by the International Pediatric Consensus Conference
3. Need for Continuous Renal Replacement Therapy (CRRT) = acute kidney injury defined by the KDIGO criteria (16) AND/OR fluid overload ≥ 10%

Exclusion Criteria:

* Refused consensus by parents
* Concomitant use of other extracorporeal blood purification techniques.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Vasopressors and inotropes reduction | 96 hours
  Proportion of patients who achieved a significant reduction in vasopressors or inotropes dose from baseline to the end of treatment.

SECONDARY OUTCOMES:
Changes in hemodynamic parameters | 96 hours
  changes in CI, SVRI, systolic pressure - Psys, diastolic pressure - Pdia, and mean pressure

OTHER OUTCOMES:
Organ dysfunction change | 96 hours
  changes in PELOD-2 score
Biomarkers of infection change | 96 hours
  time-course of C-Reactive Protein, procalcitonin
Perfusion indexes change | 96 hours
  Change lactate, PCO2 gap baseline
Mortality | 90 days
  Mortality at 28 days, at PICU and hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriella Bottari, Rome, Italy

REFERENCES:
- [Derived] Bottari G, Guzzo I, Cappoli A, Labbadia R, Perdichizzi S, Serpe C, Creteur J, Cecchetti C, Taccone FS. Impact of CytoSorb and CKRT on hemodynamics in pediatric patients with septic shock: the PedCyto study. Front Pediatr. 2023 Sep 15;11:1259384. doi: 10.3389/fped.2023.1259384. eCollection 2023. PMID 37780052